CLINICAL TRIAL: NCT00768183
Title: Phase 1, Single-Center, Open-label, Drug Interaction Study to Evaluate the Effect of Alcohol on the PK of Morphine Sulfate ER (KADIAN) Capsules in Healthy Adults Under Fasting and Fed Conditions and Relative BA to Morphine Solution
Brief Title: Comparison of KADIAN 100 mg When Dosed With Alcohol Under Fasting and Fed Conditions Compared to Water
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AA33687
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: KADIAN; morphine; alcohol; water; solution; fed; fasting
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency; Fasting | interventions — Morphine; Ethanol; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regimen A (Experimental): KADIAN Capsule + alcohol (under fasting conditions)
  Interventions: Drug: KADIAN Capsule + alcohol (under fasting conditions)
- Regimen B (Experimental): KADIAN Capsule + alcohol (under fed conditions)
  Interventions: Drug: KADIAN Capsule + alcohol (under fed conditions)
- Regimen C (Experimental): KADIAN Capsule + water (under fasting conditions)
  Interventions: Drug: KADIAN Capsule + water (under fasting conditions)
- Regimen D (Experimental): Morphine sulfate IR oral solution + water (under fasting conditions)
  Interventions: Drug: morphine sulfate IR oral solution + water

INTERVENTIONS:
Drug: KADIAN Capsule + alcohol (under fasting conditions) — Capsules 100 mg + 240 mL 40% ethanol in 4 shots of 60 mL
  Other Names: Kadian
  Arms: Regimen A
Drug: KADIAN Capsule + water (under fasting conditions) — Capsules 100mg + 240 mL in 4 shots of 60 mL
  Other Names: Kadian
  Arms: Regimen C
Drug: morphine sulfate IR oral solution + water — Morphine sulfate IR oral solution + water (under fasting conditions)
  Other Names: Morphine sulfate
  Arms: Regimen D
Drug: KADIAN Capsule + alcohol (under fed conditions) — Capsules 100 mg + 240 mL 40% ethanol in 4 shots of 60 mL
  Other Names: Kadian
  Arms: Regimen B

SUMMARY:
The objective of this study was to compare the single-dose relative bioavailability of Alpharma Branded Products Division Inc. (KADIAN) 100 mg morphine sulfate extended-release capsules when dosed with alcohol under fasting and fed conditions compared to water.

DETAILED DESCRIPTION:
This study was to evaluate the effect of consumming alcohol on the pharmacokie and bioavailability of Alpharma Branded Products Division Inc. (KADIAN) 100 mg morphine sulfate extended-release capsules under fasting and fed conditions.

In addition, the pharmacokinetics of an immediate release solution following a 20 mg dose was assessed for informational purposes and for possible modeling.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male volunteers, 21 to 40 years of age.
* Subjects were non-smokers for at least 3 months or light smokers (less than 10 pack-years).
* Subjects with a history of moderate consumption of at least 7-21 units of alcohol per week or the alcohol equivalent (12 oz beer = 5 oz of 80-proof distilled spirits = 1 unit).
* Weighing at least 70 kg and within 20% of their ideal weights (table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983).
* Medically healthy subjects with no clinically significant abnormalities in their laboratory profile and ECGs, as deemed by the Principal Investigator.
* Voluntarily consented to participate in the study.

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* In addition, history or presence of: alcoholism or drug abuse; asthma or other chronic respiratory illness; diabetes; gastrointestinal dysmotility, irritable bowel syndrome, chronic constipation or recent enteritis; hypersensitivity or idiosyncratic reaction to morphine or other opioids; hypersensitivity or idiosyncratic reaction to naltrexone, naloxone, or other opioids antagonists.
* History of no alcohol intake (alcohol-naive) or less than moderate alcohol intake.
* Subject with a history of alcohol intake exceeding the equivalence of 21 units/week or exceeding the average of 3 drinks per day.
* Subjects who had a surgery of the gastrointestinal tract (except appendectomy) which would interfere with absorption of the study drug.
* Subjects who received hepatic enzyme inducing drugs (e.g. Nizoral, Tagamet) within the previous three months.
* Subjects whose QTc interval was >450 msec at screening and prior to dosing.
* Subjects whose sitting blood pressure was less than 110/45 mm Hg at screening or 100/45 mm Hg before dosing.
* Subjects who had been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.
* Subjects who had made any significant donation or loss of blood within 56 days.
* Subjects who had made a plasma donation within 7 days prior to the study.
* Subjects with hemoglobin less than 12.0 g/dL.
* Subjects who had participated in another clinical trial within 28 days prior to the first dose.
* Subjects who had a positive urine test for drugs of abuse or alcohol.
* Subjects who had a positive test for, or had been treated for hepatitis B, hepatitis C or HIV.

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of alcohol ingestion on the pharmacokinetics of KADIAN | up to 48 hours post dosing

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics assessment of an immediate release morphine solution following a 20 mg dose | up to 24 hours post dosing

CONTACTS AND LOCATIONS:
Overall Officials: James C Kisicki, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States

REFERENCES:
- [Result] Johnson F, Wagner G, Sun S, Stauffer J. Effect of concomitant ingestion of alcohol on the in vivo pharmacokinetics of KADIAN (morphine sulfate extended-release) capsules. J Pain. 2008 Apr;9(4):330-6. doi: 10.1016/j.jpain.2007.11.009. Epub 2008 Jan 16. PMID 18201934